CLINICAL TRIAL: NCT04197323
Title: Alprostadil Liposomes for Injection for Lower Extremity Arteriosclerosis Obliteran of Phase II Clinical Trial
Brief Title: Alprostadil Liposomes for Injection for Lower Extremity Arteriosclerosis Obliteran
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QLDE201901/PRO
Record Dates: First submitted 2019-12-11; First posted 2019-12-13 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alprostadil liposomes for injection (Experimental)
  Interventions: Drug: Alprostadil liposomes for injection
- KAISHI for injection (Active Comparator)
  Interventions: Drug: Alprostadil liposomes for injection

INTERVENTIONS:
Drug: Alprostadil liposomes for injection — 40ug,once a day,continuous administration for 2 weeks

SUMMARY:
This is a randomized, positive-control, multicenter, multiple-dose, dose-escalation phase II trial

DETAILED DESCRIPTION:
A randomized, positive-control, multicenter, multiple-dose, dose-escalation phase II trial. The trial was divided into 4 dose groups: the positive drug Kaishi 10 μg group and the alprostadil liposome for injection 40μg, 80μg, 120μg group.

ELIGIBILITY:
Inclusion Criteria:

1. 40 <age ≤ 80 years ，regardless of gender;
2. Agree to participate in this clinical trial and sign the informed consent voluntarily;
3. Meet the diagnostic criteria of lower extremity arteriosclerosis obliteran (lower extremity ASO) (according to the definition of the 2015 Chinese lower extremity arteriosclerosis obliteran diagnosis and treatment guidelines), which are: age> 40 years; have clinical manifestations of lower extremity arteriosclerosis obliteran ; Weakness or disappearance of distal arterial pulsation in ischemic limbs;
4. Ankle-brachial index (ABI) <0.9;
5. Fontaine stage II or III. For subjects with Fontaine stage II, intermittent claudication distance is between 50m and 800m (fixed plate speed 3km / h, slope 12%); and at least 2 tests with difference of ≤25% (comparison based on the first measurement value, the second measurement is performed after the subject is fully rested the next day and after);
6. Imaging examinations such as color Doppler ultrasound, CTA, MRA, or DSA within 1 month before enrollment revealed lesions such as stenosis or occlusion of the corresponding lower limb arteries.

Exclusion Criteria:

1. Patients with pre-existing cardiac dysfunction, such as untreated heart failure, arrhythmia, coronary heart disease, mitral or aortic stenosis, or a history of myocardial infarction within the last 6 months;
2. Combining a history of stroke or cerebral hemorrhage, the judgment of researchers will affect the safety evaluation of efficacy;
3. Patients diagnosed or suspected of having pulmonary edema, pulmonary infiltration, or interstitial pneumonia through clinical or related examinations, or those with severe chronic obstructive ventilation disorder or respiratory insufficiency;
4. Obesity (BMI≥40);
5. Fontaine stage is IV, or patients with severe resting pain need to use strong analgesics or surgical amputation;
6. Hepatic impairment (ALT or AST ≥ 3 times ULN) or primary liver disease;
7. Renal dysfunction, SCr> 1.5 times the upper limit of normal value;
8. Poorly controlled hypertension (systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥110 mmHg);
9. Diabetic patients with poor control (HbA1c> 9%);
10. Patients with a history of interventional or bypass surgery or endovascular treatment in the past 3 months; or those who have stopped using prostaglandins for less than 5 half-life of the corresponding drugs; Elderly within 5 half-life of the corresponding drug (such as naphthylamine, pentoxifylline, butrodil, cilostazol, etc.);
11. Patients who have successfully received walking rehabilitation training in the past 6 months;
12. There are other diseases that significantly affect the walking distance, such as lower extremity joint disease, spinal disease, neuropathyt;
13. Patients with inflammatory vascular diseases, such as multiple arteritis, peripheral edema, thrombo-occlusive vasculitis, etc .;
14. Patients with total femoral or above, femoropopliteal artery occlusion, or above groin artery occlusion;
15. Patients with active peptic ulcer or bleeding tendency;
16. Glaucoma or hypertensive patients;
17. Patients who have used powerful analgesics (such as morphine) in the nearly a month;
18. Patients with mental illness or dementia;
19. Patients with malignant tumors;
20. Patients with previous allergies to similar products;
21. Those who have participated in drug clinical trials in the past 3 months;
22. Patients who are pregnant or nursing, or patients who are unable to perform effective contraception during the study period;
23. Active hepatitis B virus infection (HBV surface antigen positive and (HBVDNA quantification ≥1 × 103copies / mL), hepatitis C virus, syphilis antibody and HIV antibody positive;
24. Other patients considered by investigators to be unsuitable for this trial.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
intermittent claudication distance | After 2 weeks of treatment
  Change of intermittent claudication distance from baseline after 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality, China